CLINICAL TRIAL: NCT04658849
Title: Insulin Resistance Following Androgen Deprivation Therapy in Men With Prostate Cancer
Brief Title: Insulin Resistance Following ADT for Prostate CA
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: End of grant funding
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Sameer Siddiqui, MD FACS, C. Rollins Hanlon Endowed Chair of Surgery, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 30509
Record Dates: First submitted 2020-10-27; First posted 2020-12-09 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Insulin Resistance; Prostate Cancer
Keywords: Androgen Deprivation Therapy
MeSH Terms: conditions — Insulin Resistance; Prostatic Neoplasms | interventions — Pioglitazone; Tablets

STUDY DESIGN:
Intervention Model Description: We plan to conduct a prospective, randomized, double-blind, placebo-controlled trial in 44 men with nonmetastatic prostate cancer who will receive ADT with long acting GnRH agonist.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pioglitazone Arm (Experimental): Subjects will self-administer a 30 mg pioglitazone oral tablet daily for 6 months.
  For patient taking a diabetic regimen of gemfibrozil, the dose will be 15 mg daily.
  Interventions: Drug: Pioglitazone 30 Mg Oral Tablet
- Placebo Arm (Placebo Comparator): Subjects will self-administer an oral placebo tablet containing cellulose daily for 6 months.
  Interventions: Drug: Pioglitazone placebo tablet

INTERVENTIONS:
Drug: Pioglitazone 30 Mg Oral Tablet — Subjects will self-administer a 30 mg pioglitazone oral tablet daily for 6 months.
  For patient taking a diabetic regimen of gemfibrozil, the dose will be 15 mg daily.
  Other Names: Actos
  Arms: Pioglitazone Arm
Drug: Pioglitazone placebo tablet — Subjects will self-administer an oral placebo tablet containing cellulose daily for 6 months.
  Other Names: Placebo
  Arms: Placebo Arm

SUMMARY:
Prostate cancer is the most common cancer in men in the United States. Suppression of male hormone levels by using GnRH agonist ("hormone blocking therapy") for a few years is routinely used to treat prostate cancer. While the treatment is very effective, it decreases muscle mass and increases fat mass. This results in a decrease in insulin action (also called insulin resistance) and increases the likelihood of diabetes. It may also contribute to risk of developing heart disease. The investigators propose to conduct a trial that will:-

1. study the mechanisms through which GnRH agonists cause insulin resistance.
2. Evaluate a treatment that can decrease insulin resistance. This is a randomized, placebo controlled, double-blind trial. Forty-four men with prostate cancer will be recruited in the trial before starting GnRH agonist therapy. Participants will undergo metabolic studies to evaluate insulin action (called insulin clamp), abdominal fat tissue biopsy to study insulin action at the cellular level and blood draws. The study volunteers will then be given either a placebo tablet or pioglitazone tablet to take once a day for the next six months. The metabolic tests, blood test and fat tissue biopsy will be obtained again at the end of the study.

DETAILED DESCRIPTION:
STUDY PLAN The Study will be conducted at Saint Louis University. The investigators plan to conduct a prospective, randomized, double-blind, placebo-controlled trial in 44 men with nonmetastatic prostate cancer who will receive ADT with long acting GnRH agonist. Patients will be recruited from clinical practice of division of Urology. The patients that are planning to undergo ADT as part of standard of care treatment for their prostate cancer will be offered a choice of enrolling in the study prior to initiating ADT.

Study subjects will undergo EHC, subcutaneous fat biopsy and have a blood sample drawn prior to starting ADT. The subjects will then be randomized to 30 mg pioglitazone or placebo tablet daily for 6 months. Blood samples will be drawn 2 and 4 months following the initiation of the study drug. The final study visit will be at 6 months. Subjects will undergo EHC, fat biopsy and blood sampling and will be discharged from the study. Study visits will be conducted at clinical research center of division of Endocrinology at Salus Center.

Screening:

All subjects will complete the following procedures prior to participating in the study:-

1. Medical History. Subjects who are on insulin or sulfonylureas for diabetes will be advised that pioglitazone use may lead to low blood sugars. Subjects with congestive heart failure will be advised of the possibility that their edema or shortness of breath may worsen.
2. Physical Exam
3. Informed consent
4. Lab test: CBC and comprehensive metabolic panel (CMP) if not available in medical records from last 3 months

Subjects who qualify and consent to take part in the study will be assigned a number by a computerized random number generation program and will be randomized (1:1) to receive either pioglitazone or placebo. An unblinded pharmacist will prepare the study product. Study investigators, staff and the study participants will be blinded.

Baseline study visit: This visit will happen prior to starting ADT. The participants will come fasting and have blood drawn to measure CBC, comprehensive metabolic panel (CMP), total and free testosterone, SHBG and LH. MNC and serum will be stored for the research laboratory. Subcutaneous fat biopsy will be performed. Following the biopsy, EHC will be started (procedures described below). Subjects will be given an 8 week supply of pioglitazone 30 mg or placebo pills containing cellulose. For patient taking gemfibrozil, the dose will be 15 mg daily. Subjects will start the study drug one week after initiating the ADT. The subjects will take the study drug once a day in the morning. Subjects who take insulin or sulfonylureas will be asked to contact their doctor and report to the study team if hypoglycemia is experienced. The study physician may change the diabetes therapy if warranted. A letter will be sent to providers (who manage patient's diabetes) of all patients notifying them of possible changes in patient's diabetes regimen. All subjects with heart failure will be advised to report shortness of breath or worsening of edema to their doctors and to the study team.

Weeks 8 and 16 study visits: The participants will come fasting and have blood drawn for research laboratory. Participants will be given supply of study drug for another 8 weeks. Participants will be seen by a study physician for physical exam. Diabetic patients using insulin or sulfonylureas will discuss their blood sugars with the study physician. The study physician may choose to decrease the dose or stop insulin or sulfonylureas to avoid hypoglycemia. If therapy is changed, a letter will be sent to patient's diabetes provider.

Week 24 study visit (end of study): The participants will come fasting and have blood drawn to measure CBC, CMP, total and free testosterone, SHBG. Blood will be drawn. MNC and serum will be stored for the research laboratory. Subcutaneous fat biopsy and EHC will be performed. The subjects will then be discharged from the study and follow with their physicians. Diabetic patients will be told of the possibility that their blood sugars may increase.

PROCEDURES Measurement of whole body glucose uptake by hyperinsulinemic euglycemic clamp: Subjects will come to the clinical research center in the morning after an overnight 10 hour fast. Patients with blood sugar >180 mg/dl will be re-scheduled. Diabetes medications will be held on the morning of EHC. Long acting insulin (if being taken) will be held the night before the clamp. Insulin clamp will be started with a priming dose of short acting human insulin given over 10 minutes and then an infusion at the rate of 80mU/m2/min. 20% glucose infusion will be started at 5 minutes and glucose infusion rate will be titrated to maintain blood glucose concentration at 90 mg/dl. Twenty mEq of KCL will be added to one liter of 20% glucose. Insulin will be infused for three hours. Blood sample will be collected to measure insulin concentrations at 0, 60, 120, 150 and 180 minutes. Insulin sensitivity will be calculated from the glucose infusion rates during the last 30 min of the clamp (steady state) divided by the steady-state plasma insulin concentration divided by body weight.

Fat aspiration procedure: Subcutaneous fat tissue aspiration will be performed on abdomen at a 10 cm distance from umbilicus. The skin will first be prepared and a sterile drape will be placed around the appropriate area. Under local anesthesia, 500mg-3g of fat tissue will be obtained. The adipose tissue will be centrifuged to remove blood and fluid contaminants. The upper adipose tissue will be collected into a separate sterile tube, washed twice with cold sterile Phosphate Buffered Saline and centrifuged to remove the saline. Total RNA, nuclear extracts and total cell lysates will be prepared from the adipose tissue.

Clinical laboratory assays: Total and free testosterone concentrations will be measured by liquid chromatography tandem mass spectrometry and equilibrium dialysis (12). SHBG, LH, CBC, CMP will be measured by standard assays. All measurements will be carried out by Quest diagnostics.

Mononuclear cells (MNC) isolation: Blood samples will be collected in Na-EDTA and carefully layered on Lympholyte medium (Cedarlane Laboratories, Hornby, ON). Samples will be centrifuged till two bands separate out at the top of the RBC pellet. The MNC band will be harvested and washed twice with Hank's balanced salt solution. This method provides yields greater than 95% MNC preparation.

Quantification of mRNA Expression by RT-PCR: Expression of inflammatory mediators involved in insulin resistance and those that mediate insulin signaling will be tested by RT-PCR in mRNA isolated from MNC and adipose tissue. Total RNA will be isolated from MNC and adipose tissue using commercially available RNAqueous®-4PCR Kit and adipose tissue RNA Isolation kit (Ambion, Austin, TX). Real Time RT-PCR will be performed using Stratagene Mx3000P QPCR System (La Jolla, CA), Sybergreen master mix(Qiagen, CA) and gene specific primers for IKK-β, SOCS-3, PTEN, PTP-IB, JNK-1, TLR-4, IL-1β, IR, IRS-1, AKT-2, GLUT-4 (Life Technologies, MD). All values will be normalized to the expression of a group of housekeeping genes including actin, ubiquitin C and cyclophilin A. The normalization factor used is calculated by GeneNorm software and is based on the values of all housekeeping genes used.

Western blotting: MNC and adipose tissue total cell lysates will be prepared. Electrophoresis and immunoblotting will be carried as described before (13). Polyclonal antibodies against IR, AKT-2, SOCS-3, IKK-β and actin will be used and all values will be corrected for loading to actin.

Plasma measurements: ELISA will be used to measure plasma concentrations of insulin, C-reactive protein, adiponectin, TNF-α and IL-1β. FFA concentrations will be measured by a colorimetric assay. The research laboratory measurements will be conducted in the Endocrine laboratory at Doisy Hall.

Data Analysis: The focus of the proposed research is to evaluate the efficacy of pioglitazone treatment on insulin sensitivity men receiving ADT. Transformations of the data in order to meet statistical assumptions may be considered. The results will be computed as mean ± standard deviation. The primary endpoint of the study is to detect a difference in insulin sensitivity as measured by whole body glucose uptake during EHC after treatment with pioglitazone as compared to placebo. There are no prior studies analyzing the effect of pioglitazone in men undergoing ADT. However, studies of pioglitazone in patients with type 2 diabetes have shown an increase in insulin sensitivity of ~30% (14-16). Change in insulin sensitivity following pioglitazone or placebo for 24 weeks will be compared among the groups by unpaired t-test. Estimating a difference in insulin sensitivity of 30%, a sample size of 22 patients per treatment group (assuming a drop-out rate of 20%) should provide adequate power (Beta = 0.8) to detect a significant difference (alpha = 0.05), provided the standard deviation of the residuals is not greater than the mean difference. Thus 44 men will be recruited in the study.

Secondary End Points: The secondary endpoints for the study will be comparison of the relative change from baseline in HOMA-IR, insulin signaling and inflammatory mediators after pioglitazone or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Men between the ages of 18-85 years
2. Prostate cancer, non-metastatic
3. Planning to initiate ADT with long acting GnRH agonist

Exclusion Criteria:

1. Prior history of ADT use
2. Used pioglitazone in last 6 months
3. Congestive Heart Failure Class 3 or 4
4. Osteoporosis, including history of fragility fracture
5. history of bladder cancer
6. Hemoglobin <8 g/dl
7. eGFR <15 ml/min/1.73m2
8. liver enzymes (ALT or AST) >3 times the upper limit of normal

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
Insulin Sensitivity | 6 months
  The primary endpoint of the study is to detect a difference in insulin sensitivity as measured by whole body glucose uptake during EHC after treatment with pioglitazone as compared to placebo.

SECONDARY OUTCOMES:
HOMA-IR | 6 months
  A secondary endpoint for the study will be comparison of the relative change from baseline in HOMA-IR after pioglitazone or placebo.
Insulin signaling | 6 months
  A secondary endpoint for the study will be comparison of the relative change from baseline in insulin signaling after pioglitazone or placebo.
C Reactive Protein | 6 months
  A secondary endpoint for the study will be comparison of the relative change from baseline in C Reactive Protein after pioglitazone or placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Sameer Siddiqui, MD, Principal Investigator — St. Louis University; Sandeep Dhindsa, MD, Study Director — St. Louis University
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No